CLINICAL TRIAL: NCT05258591
Title: Portable Method of Motor Rehabilitation Using Functional Near-InfraRed Spectroscopy- Based Brain-computer-interface to Augment Post-stroke Recovery (fNIRS-PROMOTE- Recovery)
Brief Title: Post-stroke Motor Rehabilitation Using Functional Near-infrared Spectroscopy-based Brain-computer-interface
Acronym: fNIRS-PROMOTE
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Axem Neurotechnology Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020A016951
Record Dates: First submitted 2022-01-18; First posted 2022-02-28 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Axem Home (Experimental): Patients receive at-home access to Axem Home system for duration of the study period.
  Interventions: Device: Axem Home

INTERVENTIONS:
Device: Axem Home — Rehabilitation system comprised of functional near-infrared spectroscopy headband (measuring from the motor cortex), as well as tablet-based software application (guiding stroke survivors through rehabilitation exercises for their hands/arms).

SUMMARY:
Chronic stroke survivors suffering from weaknesses or movement difficulties in their hand/arm are provided a system to aid in at-home rehabilitation for 6 weeks. This rehabilitation system includes a headband that measures and provides feedback from the brain during rehabilitation, together with tablet-based software. Throughout the 6 week rehabilitation period (as well as in a follow-up session 1 month afterwards) several assessments are taken to understand the effect of this rehabilitation on participant's movement abilities, as well as their brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 90 years
* 6 months - 5 years since most recent stroke
* Upper-extremity Fugl-Meyer motor function (FMA-UE) score ≤56
* Able to follow simple commands
* Fluency in English
* Not currently receiving therapy for the upper extremity

Exclusion Criteria:

* Visual impairment that would interfere with visualization of the therapy interface (score >0 on the visual subscale of the NIH stroke scale)
* Montreal Cognitive Assessment (MoCA) Score ≥10
* History of significant physical disability prior to most recent stroke
* Open wounds on the scalp
* Unable or unwilling to remove hair braids or head coverings which interfere with the Axem Home device efficacy.
* Inability to follow training instructions for at-home BCI system.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Determine whether there are participants who respond to at-home upper-extremity BCI rehabilitation. | 6 weeks
  Some participants will demonstrate a pre- to post-test increase of 6 in the Fugl-Meyer Upper-Extremity subscale.
Determine whether there are participants who respond to at-home upper-extremity BCI rehabilitation. | 6 weeks
  Some participants will demonstrate a pre- to post-test increase of 12 in the Action Research Arm Test.
Determine whether there are participants who respond to at-home upper-extremity BCI rehabilitation. | 6 weeks
  Some participants will demonstrate a pre- to post-test increase of either 0.5 in the Motor Activity Log.
Determine whether there are participants who respond to at-home upper-extremity BCI rehabilitation. | 6 weeks
  Some participants will demonstrate a pre- to post-test minimally clinically important differences the Stroke Impact Scale.
Determine when in the course of the study (if at all) fNIRS data contains predictive information regarding the likelihood that participants would respond to at-home BCI rehabilitation. | 6 weeks
  Significant differences between responders and non-responders (as defined in the endpoint of primary objective 1) in fNIRS measures taken either during pre-test fNIRS tasks or at-home BCI sessions which are not accounted for by pre-test FMA-UE assessment scores (see Statistical Methods below for more information).
Determine when in the course of the study (if at all) fNIRS data contains predictive information regarding the likelihood that participants would respond to at-home BCI rehabilitation. | 6 weeks
  Significant differences between responders and non-responders (as defined in the endpoint of primary objective 1) in fNIRS measures taken either during pre-test fNIRS tasks or at-home BCI sessions which are not accounted for by pre-test ARAT assessment scores (see Statistical Methods below for more information).

SECONDARY OUTCOMES:
Determine whether participants can learn to modulate motor cortex brain activity during at-home BCI rehabilitation using a prototype wireless fNIRS device. | 6 weeks
  A significant difference between mean ∆HbO during either (1) the MI Task conducted at the pre-test period and MI during at-home BCI sessions conducted during week 5 and/or (2) the Motor Execution Task conducted at the pre-test ME Task and ME during at-home BCI sessions conducted during week 5 (see Statistical Methods below for more information).
If secondary objective 1 is met, determine whether learning to modulate motor cortex brain activity during at-home BCI rehabilitation increases the likelihood of benefitting from at-home BCI rehabilitation. | 6 weeks
  A significant relationship between the ability to modulate motor cortex brain activity during at-home BCI (as defined in the endpoint of secondary objective 1) and their change in FMA-UE from their pre- to post-test assessments (see Statistical Methods below for more information).
If secondary objective 1 is met, determine whether learning to modulate motor cortex brain activity during at-home BCI rehabilitation increases the likelihood of benefitting from at-home BCI rehabilitation. | 6 weeks
  A significant relationship between the ability to modulate motor cortex brain activity during at-home BCI (as defined in the endpoint of secondary objective 1) and their change in ARAT from their pre- to post-test assessments (see Statistical Methods below for more information).
If any of primary objectives 1-4 are met, show that the improvements in function achieved by responders to at-home BCI rehabilitation is maintained after the at-home BCI rehabilitation is discontinued. | 10 weeks
  At least one of the significant differences in FMA-UE scores observed between the pre- and post-tests are maintained at the follow-up session (see Statistical Methods below for more information).
If any of primary objectives 1-4 are met, show that the improvements in function achieved by responders to at-home BCI rehabilitation is maintained after the at-home BCI rehabilitation is discontinued. | 10 weeks
  At least one of the significant differences in ARAT scores observed between the pre- and post-tests are maintained at the follow-up session (see Statistical Methods below for more information).

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States